CLINICAL TRIAL: NCT02874443
Title: The REDUCED Trial: REDucing the Utilization of CEsarean Sections for Dystocia
Acronym: REDUCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Stephen Wood, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB16-1576
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section, Dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention centers (Experimental): Application of a knowledge translation strategy, of new clinical practice guidelines on labor management, to physicians and nurses caring for women in labor.
  Intervention centers will receive knowledge translation of labor management guidelines
  Interventions: Other: Knowledge Translation of labor management guidelines
- Control centers (No Intervention): No intervention at control centers

INTERVENTIONS:
Other: Knowledge Translation of labor management guidelines
  Arms: Intervention centers

SUMMARY:
This project is a clustered randomized controlled trial of a knowledge translation intervention of new ACOG guidelines for the diagnosis of poor progress in labor. The intent is to reduce the rate of cesarean section (CS) in first time mothers at term (>= 37 weeks), with a vertex presenting singleton fetus, without increasing maternal or neonatal morbidity. The guidelines were developed from data from the Consortium for Safe Labor. The unit of randomization will be sites in Alberta that deliver

DETAILED DESCRIPTION:
Cluster randomized controlled trial of a knowledge translation intervention of new guidelines for the diagnosis of poor progress in labor. The intervention will be randomized to centres (the clusters) in Alberta that provide intrapartum care, have facilities to perform cesarean section and deliver at least 70 primparous women annually, with stratification based on facility type and geographic location. Clustering by centre and not individual caregivers (nurses/physicians) is necessary to prevent leakage or crossover of the intervention to controls. As all participating centres will eventually receive the intervention, the biostatistician will generate a randomization into two "waves". The intervention will be introduced sequentially by strata (Calgary, Edmonton, regional centres, rural centres) to the first "wave" hospitals in multi-week run-in periods after which those strata will be revisited for roll-out to the second "wave" hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Centers in Alberta that provide intrapartum care, have facilities to perform cesarean section and deliver at least 70 primparous women annually

Exclusion Criteria:

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88918 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Rate of Cesarean section | at delivery
  Rate of Cesarean section in primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus

SECONDARY OUTCOMES:
Rate of perinatal death | at delivery
  Rate of perinatal death for primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of neonatal asphyxia | at delivery
  Neonatal asphyxia is defined as intrapartum stillbirth or neonatal death from asphyxia (Perinatal Society of Australia and New Zealand coding) or Neonatal Intensive Care Unit admission and at least two of: a. Apgar score of ≤5 at 10 minutes; b. Mechanical ventilation or chest compressions for resuscitation within 10 minutes; c. Cord pH < 7.00 (venous or arterial), or arterial base excess ≥ 12 at birth. Rate of neonatal asphyxia for deliveries involving primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of moderate or severe asphyxia or meets criteria for therapeutic cooling | at delivery
  Rate of moderate or severe asphyxia or meets criteria for therapeutic cooling for deliveries involving primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of neonatal sepsis or suspected sepsis | at delivery
  Rate of neonatal sepsis or suspected sepsis for deliveries involving primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of post partum hemorrhage | at delivery
  Rate of post partum hemorrhage for primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of blood transfusion | at delivery
  Rate of blood transfusion for primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of postpartum uterine artery/pelvic artery embolization | Within 30 days of delivery
  Rate of postpartum uterine artery/pelvic artery embolization for primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of postpartum hysterectomy | Within 30 days of delivery
  Rate of postpartum hysterectomy for primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus
Rate of postpartum maternal intensive care unit (ICU) admission | at delivery
  Rate of postpartum maternal intensive care unit (ICU) admission for primiparous women in labor, at term (>= 37 weeks), with a vertex presenting singleton fetus

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Wood, MD MSc, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Wood S, Skiffington J, Brant R, Crawford S, Hicks M, Mohammad K, Mrklas KJ, Tang S, Metcalfe A; REDUCED Trial Team. The REDUCED trial: a cluster randomized trial for REDucing the utilization of CEsarean delivery for dystocia. Am J Obstet Gynecol. 2023 May;228(5S):S1095-S1103. doi: 10.1016/j.ajog.2022.10.038. Epub 2023 Mar 16. PMID 37164490

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/43/NCT02874443/Prot_SAP_007.pdf